CLINICAL TRIAL: NCT02358486
Title: Effect and Mechanism of Acupuncture on Patients With Functional Dyspepsia: a Protocol for a Randomized, Assessor-blind, Sham-controlled Trial
Brief Title: The Effect and Mechanism of Acupuncture on Functional Dyspepsia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government); Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Seok-Jae Ko, PhD, Professor, Department of Korean Internal Medicine, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KHNMCOH 2014-08-002
Record Dates: First submitted 2015-01-21; First posted 2015-02-09 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Dyspepsia
Keywords: Functional Dyspepsia; Acupuncture; Functional MRI
MeSH Terms: conditions — Dyspepsia | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acupuncture (Experimental): Participants in this group are given 10 times of real acupuncture treatment for 4 weeks.
  Interventions: Device: Acupuncture
- Sham acupuncture (Sham Comparator): Participants in this group are given 10 times of sham acupuncture treatment for 4 weeks.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Acupuncture — 1. Acupuncture rationale 1a) Style of acupuncture: body acupuncture (in accordance with meridian theory)
  2. Needling details 2a) Number of needle insertions per subject per session: 13 2b) Acupoints: Basic points - Large Intestine(LI)4, Stomach(ST)36, Liver(LR)3, Pericardium(PC)3, Spleen(SP)4, Stomach(ST)34, Conception Vessel(CV)12, 2c) Depth: 5 ~ 30mm 2d) Response sought: 'De qi' sensation; 2e) Needle stimulation: Manipulation 2f) Retention time: 15 minutes 2g) Needle type: 0.2 X 40 mm, sterilized stainless steel needle, Dongbang Inc., Korea
  Other Names: Acupuncture treatment
  Arms: Acupuncture
Device: Sham acupuncture — The participants in sham acupuncture group are given sham acupuncture treatment at the same acupoints in the same times and method as acupuncture arm. The sham device would be a Streitberger device.
  Other Names: Streitberger Device
  Arms: Sham acupuncture

SUMMARY:
The aim of the study is to investigate the effect of acupuncture on functional dyspepsia compared with sham control. The study aims to clarify the mechanism of acupuncture by assessing functional magnetic resonance imaging and metabolomics.

DETAILED DESCRIPTION:
Functional dyspepsia (FD) is a functional gastrointestinal disorder without any structural lesion. Due to the lack of satisfactory effect of conventional treatments, many FD patients turn to alternative treatments such as acupuncture. Acupuncture, one of the most sought therapeutic modalities in traditional Korean Medicine, has been commonly used for treating gastrointestinal disorders.

However, the effect and mechanism of acupuncture on FD has not been rigorously evaluated. In the present study, we will investigate whether 10 sessions of acupuncture over 4 weeks, in comparison with sham acupuncture, improve symptoms of FD and activate regions of brain area. We will also perform metabolomics study to find the mechanism of acupuncture to FD. Outcome measures include proportion of responder, Korean version of Nepean Dyspepsia Index, Functional Dyspepsia-Related Quality of Life, Ways of Coping Question, Coping Strategy Questionnaire, Perception of bodily sensation, The State-Trait Anxiety Inventory, Center for Epidemiologic Studies Depression Scale, functional magnetic resonance imaging and metabolomic study.

ELIGIBILITY:
Inclusion criteria

Participants should meet following conditions:

1. Aged of 30 - 49
2. Individuals who meet FD and postprandial distress syndrome (PDS) criteria in Rome III
3. Individuals who complain the degree of dyspepsia for more than 40 points of visual analogue scale (VAS; 0, no symptom at all; 100, the most severe symptom one ever had)
4. At least 3 questions show more than 2 points in Gastrointestinal impact scale
5. Individuals who have normal esophagogastroduodenoscopy results within a year and no organic diseases which can explain current symptoms such as peptic ulcer, dysplasia, mucosa-associated, lymphoid tissue lymphoma, esophageal cancer, gastric cancer
6. Individuals who are not supposed to take any other treatments associated with FD during the study
7. Individuals who voluntarily agree with a study protocol and sign a written informed consent

Exclusion Criteria

Participants who report the followings will be excluded:

1. Individuals who have organic diseases such as gastroesophageal reflux disease
2. Individuals who have obvious signs of irritable bowel syndrome
3. Individuals who have alarm symptoms (weight loss, black or tar stool or dysphagia)
4. Individuals who have serious structural disease (disease of heart, lung, liver or kidney) or mental illness
5. Individuals who have had surgery related with the gastrointestinal tract , except for appendectomy more than six months ago
6. Individuals who are pregnant or breastfeeding
7. Individuals who are taking drugs which might affect gastrointestinal tract; minimum wash-out period of 2 weeks is required before participating in the trial
8. Individuals who are HIV-positive
9. Individuals who have a problem of mal-absorption
10. Individuals who have difficulties in attending the trial (eg. paralysis, serious mental illness, dementia, drug addiction, time constraint, severe disorder in vision or hearing, illiteracy, etc.)
11. Individuals who do not want to sign the informed consent
12. Individuals who have other diseases that could interfere acupuncture treatment, e.g. clotting disorders or leukopenia, pace-maker, epilepsy, or anticoagulant therapy
13. Individuals who have metal implants or fragments which might influence fMRI examination

Ages: 30 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of responders | Once in treatment period (4 wks)
  The proportion of patients who answer "Yes" to more than half of adequate relief questions in the treatment period. Patients are expected to report their response to the acupuncture treatment by answering the following question at each visit: "After the last visit, have you had adequate relief of your stomach pain or discomfort?" Questions will be asked at each visit during treatment period (Twice a week for 4 wks, total 10 times - 0, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 4.5 wks). Responders are defined as patients reporting adequate relief for at least 50% of the study period (more than 5 times of "Yes" to adequate relief question out of total 10 questions). The proportion of responder will be compared statistically between intervention groups.

SECONDARY OUTCOMES:
Nepean Dyspepsia Index - Korean version (NDI-K) | treatment (0 wks), After treatment (4 wks)
  The Nepean Dyspepsia Index is a reliable and valid measure of quality of life in FD. The Nepean Dyspepsia Index originally contains 42 items designed to measure impairment of a subjective ability engaged in relevant aspects of their life because of dyspepsia. It was subsequently shortened to 25 items, yielding 5 sub-scales. NDI-K, validated in 2003 by Lee at al., made up of 2 sections which are about symptom-based questions and quality of life. In this trial, symptom-based questions, i.e. questions about period, severity and distressful degree of 15 symptoms, will be evaluated.
Functional Dyspepsia-Related Quality of Life (FD-QoL) Questionnaire | Before treatment (0 wks), After treatment (4 wks)
  The FD-QoL scale is a 21-item Likert-type questionnaire that can easily be completed within 5 min. Short administration time and high comprehensibility supports the feasibility of measuring health-related quality of life.
Ways of Coping Question (WCQ) | treatment (0 wks), After treatment (4 wks)
  The Ways of Coping Questionnaire (WCQ) (Folkman & Lazarus, 1988) assessed the parents' coping strategies. It has 66-items, each with a 4-point Likert scale indicating the frequency with which the strategy was used. The measure comprises eight scales representing theoretically different coping strategies: confrontative coping, distancing, self-controlling, seeking social support, accepting responsibility, escape-avoidance, problem solving, and positive reappraisal.
Coping Strategy Questionnaire (CSQ) | Before treatment (0 wks), After treatment (4 wks)
  Coping Strategy questionnaire is one of models for measuring stress and coping to help explain the differences in adjustment found among persons who experience chronic pain. It consists of 48 items, each with a 7-point Likert scale (0:never; 3: sometimes; 6:always) and divide into eight scales of six items each; (1) Catastrophizing, (2) Distractor behaviors, (3) Self-instructions, (4) Ignoring the pain, (5) Reinterpreting the pain, (6) Hoping, (7) Faith and praying, (8) Cognitive distraction.
Functional Magnetic Resonance Imaging ; 3.0T MRI system(Achieva, Philips) | Before treatment (0 wks), After treatment (4 wks)
  A measure of steady state (REST and PAIN) and blood oxygenation level dependent (BOLD) under the condition of event related design (ACUP) scan run.
Metabolic profiling of plasma and urine | Time Frame: Before treatment (0 wks), After treatment (4 wks)
  In order to investigate the biological effects of FD and the effect of acupuncture on metabolism, the blood and urine sample will be analyzed using nuclear magnetic resonance (NMR)-based metabolomic techniques to compare the metabolites such as amino acids, organic acids, and blood sugar of FD patients.
The Center for Epidemiologic Studies Depression Scale (CES-D) | Before treatment (0 wks), After treatment (4 wks)
  The Center for Epidemiological Studies-Depression (CES-D), originally published by Radloff in 1977, is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or little of the time, 2 = Moderately or much of the time, 3 = Most or almost all the time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
The State-Trait Anxiety Inventory (STAI) | Before treatment (0 wks), After treatment (4 wks)
  The State-Trait Anxiety Inventory (STAI) is a psychological inventory based on a 4-point Likert scale and consists of 40 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety (anxiety triggered by a specific event), and trait anxiety (anxiety derived from personal characteristic). Higher scores are positively correlated with higher levels of anxiety.
Perception of bodily sensation (PDS) | Before treatment (0 wks)
  This scale is a 10-item questionnaire with 6(1-7) point Likert scale. Patients with higher Perception of bodily sensation (PBS) could have a higher emotional or cognitive intolerance to bodily reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Seok-Jae Ko, KMD, PhD, Principal Investigator — Kyung Hee University Hospital at Gangdong
Locations (1):
- Kyung Hee University Hospital at Gangdong, Seoul, Gangdong-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Drossman DA. The functional gastrointestinal disorders and the Rome III process. Gastroenterology. 2006 Apr;130(5):1377-90. doi: 10.1053/j.gastro.2006.03.008. No abstract available. PMID 16678553
- [Background] Park YC, Kang W, Choi SM, Son CG. Evaluation of manual acupuncture at classical and nondefined points for treatment of functional dyspepsia: a randomized-controlled trial. J Altern Complement Med. 2009 Aug;15(8):879-84. doi: 10.1089/acm.2008.0369. PMID 19678778
- [Background] Park HJ, Kim ST, Yoon DH, Jin SH, Lee SJ, Lee HJ, Lim S. The association between the DRD2 TaqI A polymorphism and smoking cessation in response to acupuncture in Koreans. J Altern Complement Med. 2005 Jun;11(3):401-5. doi: 10.1089/acm.2005.11.401. PMID 15992222
- [Background] Talley NJ, Locke GR 3rd, Herrick LM, Silvernail VM, Prather CM, Lacy BE, DiBaise JK, Howden CW, Brenner DM, Bouras EP, El-Serag HB, Abraham BP, Moayyedi P, Zinsmeister AR. Functional Dyspepsia Treatment Trial (FDTT): a double-blind, randomized, placebo-controlled trial of antidepressants in functional dyspepsia, evaluating symptoms, psychopathology, pathophysiology and pharmacogenetics. Contemp Clin Trials. 2012 May;33(3):523-33. doi: 10.1016/j.cct.2012.02.002. Epub 2012 Feb 10. PMID 22343090
- [Background] Kaptchuk TJ, Kelley JM, Conboy LA, Davis RB, Kerr CE, Jacobson EE, Kirsch I, Schyner RN, Nam BH, Nguyen LT, Park M, Rivers AL, McManus C, Kokkotou E, Drossman DA, Goldman P, Lembo AJ. Components of placebo effect: randomised controlled trial in patients with irritable bowel syndrome. BMJ. 2008 May 3;336(7651):999-1003. doi: 10.1136/bmj.39524.439618.25. Epub 2008 Apr 3. PMID 18390493
- [Background] Zaslawski CJ, Cobbin D, Lidums E, Petocz P. The impact of site specificity and needle manipulation on changes to pain pressure threshold following manual acupuncture: a controlled study. Complement Ther Med. 2003 Mar;11(1):11-21. doi: 10.1016/s0965-2299(02)00116-4. PMID 12667970
- [Background] Park JW, Ko SJ, Han G, Yeo I, Ryu B, Kim J. The Effects of Banha-sasim-tang on Dyspeptic Symptoms and Gastric Motility in Cases of Functional Dyspepsia: A Randomized, Double-Blind, Placebo-Controlled, and Two-Center Trial. Evid Based Complement Alternat Med. 2013;2013:265035. doi: 10.1155/2013/265035. Epub 2013 Jun 3. PMID 23861702
- [Background] Labus JS, Gupta A, Coveleskie K, Tillisch K, Kilpatrick L, Jarcho J, Feier N, Bueller J, Stains J, Smith S, Suyenobu B, Naliboff B, Mayer EA. Sex differences in emotion-related cognitive processes in irritable bowel syndrome and healthy control subjects. Pain. 2013 Oct;154(10):2088-2099. doi: 10.1016/j.pain.2013.06.024. Epub 2013 Jun 20. PMID 23791896
- [Background] Rodriguez Franco L, Cano Garcia FJ, Blanco Picabia A. [Assessment of chronic pain coping strategies]. Actas Esp Psiquiatr. 2004 Mar-Apr;32(2):82-91. Spanish. PMID 15042468
- [Background] De Giorgi F, Sarnelli G, Cirillo C, Savino IG, Turco F, Nardone G, Rocco A, Cuomo R. Increased severity of dyspeptic symptoms related to mental stress is associated with sympathetic hyperactivity and enhanced endocrine response in patients with postprandial distress syndrome. Neurogastroenterol Motil. 2013 Jan;25(1):31-8.e2-3. doi: 10.1111/nmo.12004. Epub 2012 Aug 21. PMID 22908903
- [Derived] Ko SJ, Park K, Kim J, Kim M, Kim JH, Lee J, Mohamed AZ, Yeo I, Kim J, Choi SM, Kim H, Park JW, Lee JH. Effect of acupuncture and its influence on cerebral activity in functional dyspepsia patients: study protocol for a randomized controlled trial. Trials. 2016 Apr 2;17:183. doi: 10.1186/s13063-016-1296-2. PMID 27039086